CLINICAL TRIAL: NCT06537063
Title: Early Diagnosis Value of G-quadruplex DNA Methylation in Patients with Cancer
Brief Title: Detection of G-quadruplex DNA Methylation in Cancer
Status: Withdrawn | Type: Observational
Why Stopped: The existing basic research and the latest literature reports do not support the proposed protocol, therefore, the project is withdrawn.
Sponsor: Zhongnan Hospital (Other)
Responsible Party: Principal Investigator, Yu Xiao, Director, Zhongnan Hospital
Other Study IDs: YX202401
Record Dates: First submitted 2024-07-31; First posted 2024-08-05 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2024-07

CONDITIONS: Cancer; DNA G-quadruplex; Methylation; Cell-free DNA
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Asymptomatic population: Asymptomatic medical examination population.
  Interventions: Other: G4 DNAm test

INTERVENTIONS:
Other: G4 DNAm test — Detection of DNA methylation (DNAm) around G-quadruplex loci in cell-free DNA from blood.

SUMMARY:
This study aims to evaluate the early diagnosis value of G-quadruplex DNA methylation in patients with cancer.

DETAILED DESCRIPTION:
Global DNA hypomethylation is a hallmark of most cancers that occurs early during oncogenesis. We would like to investigate whether cancer-specific transcription factor binding to DNA G-quadruplex drives DNA hypomethylation in cancer. In this observational study, we would like to clarify whether DNA hypomethylation around G-quadruplex loci in cell-free DNA could be detected in early-stage cancer patients from healthy donors with high sensitivity and specificity.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers identified as asymptomatic during medical examination;
* Age≥42 years old;
* Voluntarily participate in this study and sign the informed consent.

Exclusion Criteria:

* History of malignancy or having achieved complete remission following tumor surgery;
* Certain autoimmune diseases (e.g., systemic lupus erythematosus, Sjögren's syndrome, antiphospholipid syndrome, rheumatoid arthritis, Crohn's disease, IgA nephropathy, myasthenia gravis, dermatomyositis, immune thrombocytopenic purpura, etc.);
* Pregnancy;
* Acute trauma (including surgical procedures), sudden onset organ failure (e.g., resulting from a car accident, fulminant hepatic failure, acute pancreatitis, severe pneumonia due to influenza virus), or diagnosis of sepsis;
* Previous receipt of allogeneic blood transfusion, transplant surgery, or allogeneic cell therapy;
* Volunteers who cannot provide informed consent.

Min Age: 42 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers, aged 42 years or older, who are asymptomatic as determined by medical examination and willing to participate voluntarily in the study with signed informed consent.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2024-04-30 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
G-quadruplex DNAm score | 2024.04.30-2024.09.30
  Detection of DNAm around G-quadruplex loci in cell-free DNA from blood.

CONTACTS AND LOCATIONS:
Locations (1):
- Hubei Locations, Wuhan, Hubei, China